

# Mycosis fungoides cutaneous T-cell lymphoma

# Protocol AC-079A501

# **PROVe**

A PROspective, observational, US-based study assessing outcomes, adverse events, treatment patterns, and quality of life in patients diagnosed with mycosis fungoides cutaneous T-cell lymphoma and treated with Valchlor®

Authors: Badri Rengarajan, Carol Zhao, Sandy Petersen-Stenger

Document type: Protocol for Non-Drug Interventional and Non-interventional

(Observational) Studies using Epidemiological Methods

Document status and

version:

Final Version 3

Date: 13 December 2016

Number of pages: 43

Document number: D-16.626

# **Confidentiality Statement**

The information contained in this document, especially unpublished data, is the property of Actelion Pharmaceuticals US, Inc. It is provided to third parties in confidence, and it is understood that this information will not be disclosed to any third party without written authorization from the data owner, as laid out in the respective agreement between the parties.

Doc No D-16.626

Version 3


# **CONTACT DETAILS**

| Sponsor (Data Owner) | Actelion Pharmaceuticals US, Inc. | |
|---|---|---|
| · | 5000 Shore | eline Court, Suite 200 |
| | South San Francisco, CA 94080 | |
| Clinical Study Leader/Project | Badri Rengarajan, MD | |
| Physician | | + 1-650-624-6946 |
| | Fax | + 1-650-243-2312 |
| | e-mail | badri.rengarajan@actelion.com |
| Observational Study Scientist | Carol Zhao | o, MS |
| | | + 1-650-808-6616 |
| | Fax | + 1-650-243-2312 |
| | e-mail | carol.zhao@actelion.com |
| Clinical Study Manager | nager Sandy Petersen-Stenger, MS | |
| | | + 1-650-243-2359 |
| | Fax | + 1-650-243-2312 |
| | e-mail | sandy.petersen@actelion.com |
| Drug Safety Physician | Roberto Co | ortes, MD |
| | | + 1-650-624-6945 |
| | Fax | + 1-866-227-5886 |
| | e-mail | roberto.cortes@actelion.com |
| Lead Principal Investigator | Ellen Kim, | MD (University of Pennsylvania) |
| | 8 | + 1-215-662-6722 |
| | e-mail | ellen.kim@uphs.upenn.edu |
| Study Biostatistician | David Min | k, MS (ICON Clinical Research) |
| | | + 1-415-371-2108 |
| | e-mail | david.mink@iconplc.com |

Epidemiology and Observational Studies AC-079A501 Version 3


# SIGNATURE PAGE FOR ACTELION PHARMACEUTICALS US, INC.

Hereinafter called Actelion

**TITLE:** A prospective, observational, US-based study assessing

outcomes, adverse events, treatment patterns, and quality of life in patients diagnosed with mycosis fungoides cutaneous

T-cell lymphoma and treated with Valchlor®

PROTOCOL NUMBER: AC-079A501

**AUTHORS:** Badri Rengarajan, Director, Medical Affairs;

Carol Zhao, Medical Affairs; Sandy Petersen-Stenger, Medical.

**REVIEWERS:** Daniel Rosenberg, Senior Director, Epidemiology;

Roberto Cortes, Drug Safety US;

Laurence Oster, Senior Director, Pharmacovigilance

Europe, EU QPPV;

Lilla Di Scala, Senior Director, Biostatistics; Isabelle Leconte, Senior Director, CDDM;

Frances Duffy-Warren, VP, Head Drug Regulatory US; Elke Hunsche, Head Global Market Access and Pricing

Scientific Committee.

NAME (TITLE) DATE SIGNATURE

Badri Rengarajan, MD

Clinical Study

Leader/Project Physician

16 DEC 2016

Muchiel Hengy


Doc No D-16.626


# INVESTIGATOR/INSTITUTION SIGNATURE PAGE

# Disease area

Mycosis fungoides cutaneous T-cell lymphoma

# Protocol number, acronym, study title, version

Protocol AC-079A501, PROVe, A prospective, observational, US-based study assessing outcomes, treatment patterns, adverse events, and quality of life in patients diagnosed with mycosis fungoides cutaneous T-cell lymphoma and treated with Valchlor<sup>®</sup>. Final Version 3.

I agree to the terms and conditions relating to this study as defined in this protocol and any other protocol-related documents.

| NAME | CITY | STATE | DATE | SIGNATURE |
|---------|------|-------|------|-----------|
| (TITLE) | | | | |


# **TABLE OF CONTENTS**

| CO | NTACT DET | TAILS | 2 |
|-----|------------|------------------------------------------------------|----|
| LIS | ST OF ABBR | EVIATIONS | 7 |
| PR | OTOCOL SY | NOPSIS AC-079A501 | 8 |
| PR | OTOCOL | | 17 |
| 1 | AMENDME | ENTS AND UPDATES (PROTOCOL HISTORY) | 17 |
| 2 | STUDY MII | LESTONES | 17 |
| 3 | RATIONAL | E AND BACKGROUND | 17 |
| 4 | RESEARCH | I QUESTION AND OBJECTIVES | 18 |
| 5 | RESEARCH | I METHODS | 19 |
| | 5.1 Stu | dy design | 19 |
| | | oulation (setting and study population) | |
| | 5.2.1 | | |
| | 5.2.2 | Exclusion criteria | |
| | 5.3 Vai | riables | |
| | 5.3.1 | Outcome definition and measures | 23 |
| | 5.3.2 | | |
| | 5.3.3 | • | |
| | 5.4 Dat | a sources | |
| | 5.5 Stu | dy size | 25 |
| | | a management | |
| | 5.6.1 | | |
| | 5.7 Dat | a analysis | 27 |
| | 5.7.1 | Analysis sets and groups | 27 |
| | 5.7.2 | Clinical characteristics | 27 |
| | 5.7.3 | Treatment and assessment patterns | 27 |
| | 5.7.4 | • | |
| | 5.7.5 | Adverse events | 28 |
| | 5.7.6 | Patient-completed questionnaires | 28 |
| | | ality control | |
| | 5.9 Dis | cussion of the study methods (including limitations) | 29 |
| 6 | PROTECTION | ON OF HUMAN SUBJECTS AND ETHICAL APPROVAL | 30 |

Epidemiology and Observational Studies AC-079A501 Version 3


Doc No D-16.626


| | 6.1 | Institutional Review Board/Independent Ethics Committee approve | al | 30 |
|---|---|---|---|---|
| | 6.2 | Patient informed consent | | .30 |
| | 6.3 | Patient confidentiality | | 30 |
| 7 | MANAG | EMENT AND REPORTING OF ADVERSE EVENTS | | .31 |
| | 7.1 | Definitions | | 31 |
| | 7.1.1 | Adverse event or adverse experience | | 31 |
| | 7.1.2 | • | | |
| | 7.1.3 | | | |
| | 7.2 | Secondary exposures, AE and SAE reporting to Actelion US I | | |
| | | Safety | _ | 33 |
| | 7.2.1 | Follow-up of SAEs | | 34 |
| | 7.3 | Reporting of pregnancy | | 34 |
| | 7.3.1 | Follow-up of pregnancy | | 35 |
| | 7.4 | Reconciliation | | |
| 8 | | OR DISSEMINATING AND COMMUNICATING STUDY RES | | |
| 10 | STUDY ( | COMMITTEE(S) | | 35 |
| 11 | REFERE | NCES | | .36 |
| | | LIST OF TABLES | | |
| Tab | ole 1 | eCRF Data Collection | | 21 |
| | | LIST OF APPENDICES | | |
| A | n am diss. A | | | 20 |
| | pendix A | Skindex-29 Questionnaire | | |
| | pendix B | Skindex-29 Scoring algorithm Visual Analog Scolo for provitus | | |
| | pendix C<br>pendix D | Visual Analog Scale for pruritus | | .41 |
| Ap | penuix D | lymphomasyndrome-type cutaneous | | 12 |
| Ap | pendix E | Mycosis fungoides/Sézary syndrome-type cutaneous | | .42 |
| | | lymphoma (CTCL QOL Scoring | | .43 |

Version 3

**Epidemiology and Observational Studies** AC-079A501


# LIST OF ABBREVIATIONS

| ADR | Adverse drug reaction |
|---|---|
| AE | Adverse event |
| BSA | |
| | Body surface area |
| CAILS | Composite Assessment of Index Lesion Severity |
| CTCL | Cutaneous T-cell lymphoma |
| DCF | Data clarification form |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| EDC | Electronic data collection |
| EOS | End of study |
| FDA | Food and Drug Administration |
| IEC | Independent Ethics Committee |
| IRB | Institutional Review Board |
| MCH | Mechlorethamine hydrochloride |
| MCN | Manufacturer's Control Number |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MF-CTCL | Mycosis fungoides cutaneous T-cell lymphoma |
| MF/SS-CTCL | Mycosis fungoides / Sézary syndrome-type cutaneous T-cell lymphoma |
| mSWAT | Modified Severity Weighted Assessment Tool |
| QOL | Quality of life |
| SAE | Serious adverse event |
| TNMB | Tumor-node-metastasis-blood |
| VAS | Visual Analogue Scale |


MF-CTCL Doc No D-16.626

# PROTOCOL SYNOPSIS AC-079A501


This abstract is a stand-alone summary of the study protocol

| TITLE | A <b>PRO</b> spective, observational, US-based study assessing outcomes, adverse events, treatment patterns, and quality of life in patients diagnosed with mycosis fungoides cutaneous T-cell lymphoma (MF-CTCL) and treated with Valchlor® |
|---|---|
| ACRONYM | PROVe |
| AUTHOR | Badri Rengarajan, Actelion Pharmaceuticals US, Inc. |
| RATIONALE<br>AND<br>BACKGROUND | Due to the rarity of mycosis fungoides cutaneous T-cell lymphoma (MF-CTCL), there is a dearth of epidemiologic data detailing the clinical course of the disease and its response to treatment. While topical treatment with mechlorethamine hydrochloride (MCH) has been used since the 1950s, prospective data describing the clinical course of MF-CTCL is limited. Valchlor gel is a new formulation of MCH (or nitrogen mustard) that has been shown to be safe and effective in a clinical trial and has been approved for Stage I MF-CTCL patients |
| | Prospective data on Valchlor are currently only available from the pivotal, randomized, controlled clinical trial with strict inclusion and exclusion criteria. Understanding real-world patient safety and tolerability, as well as compliance and discontinuation rates, will assist with the management of Valchlor-treated MF-CTCL patients. This study will build and extend on the data from the Valchlor clinical development program, increase the understanding of the use of Valchlor in patients with MF-CTCL and, while limited to patients treated with Valchlor, will represent the largest prospective study with any given MF-CTCL treatment. |
| | This large, non-interventional study will provide information on the use of Valchlor in a 'real-world' clinical practice setting, and increase understanding of the management and outcomes of Valchlor-treated MF-CTCL patients. Data collected includes, but is not limited to: outcomes (e.g., clinical status and healthcare utilization [MF-CTCL-related hospitalizations and emergency room visits]), adverse events (AEs; e.g., dermatitis), clinical characteristics, and treatment patterns. Finally, this study will document disease burden (e.g., pruritus) of MF-CTCL in a real-life |


MF-CTCL Doc No D-16.626


setting by collecting patient-completed symptoms and quality of life (QOL) questionnaires for patients with skin disease. The QOL tools include VAS, Skindex-29 and a newly validated Mycosis fungoides / Sézary syndrome-type cutaneous T-cell lymphoma (MF/SS-CTCL) questionnaires. RESEARCH The objectives of this study are: **OUESTION AND** To describe clinical characteristics of patients treated with **OBJECTIVES** Valchlor at enrollment and during the study observation period. To describe treatment and response assessment patterns of patients with MF-CTCL treated with Valchlor at enrollment and during the study observation period. To assess outcomes (e.g., clinical status and rates of healthcare utilization [MF-CTCL-related hospitalizations and emergency room visits]) in patients with MF-CTCL treated with Valchlor during the study observation period. To collect and describe the incidence of AEs/serious adverse events (SAEs) in patients with MF-CTCL treated with Valchlor: o To estimate the incidence of dermatitis in patients using Valchlor during the study observation period. o To describe the management of dermatitis in patients using Valchlor at enrollment and during the study observation period. To collect patient-completed and OOL symptoms questionnaires. STUDY DESIGN This is a multi-center, prospective, observational, US-based drug study. All consecutive MF-CTCL patients being treated with Valchlor will be invited to enroll in this study. Patients will undergo clinical assessments and receive standard medical care, as determined by the patients' physician, in the real-world setting. With the exception of protocol-required patient-completed questionnaires for symptoms and QOL, there are no specific or mandated clinical assessments to be performed, and patients will not receive experimental intervention or treatment as a consequence of their participation in this study.

Patients will be followed prospectively for a maximum of 2 years


MF-CTCL Doc No D-16.626


from the date of signed informed consent (enrollment) until end of study, which includes withdrawal of consent, loss to follow-up, death, or study completion. Continuation in the study is not contingent on continuation of Valchlor.

Patients currently enrolled and ongoing or newly enrolled will be offered to participate in the 24-month study of this protocol Amendment 1. Patients who enrolled under the original protocol (prior to Amendment 1) and are still ongoing in the study will be re-consented and to follow data collection specified in Table 1 of this protocol for a total of 24 months from original consent date. Patients who enrolled and have completed 1 year of the study under the original protocol will not be re-consented under Amendment 1.

# POPULATION (SETTING AND STUDY POPULATION)

This study will enroll approximately 300 consecutive patients diagnosed with MF-CTCL and being treated with Valchlor, regardless of other MF-CTCL therapies received before or at enrollment. Patients will be enrolled from up to 50 participating centers/clinics in university-affiliated or community hospitals in the US. The participation of physicians and patients in the study is on a voluntary basis.

### Inclusion criteria:

- All adult patients (≥ 18 years of age) diagnosed with MF-CTCL and being treated with Valchlor. This includes patients newly initiating Valchlor OR patients continuing treatment with Valchlor:
  - o Patients newly initiating Valchlor are patients who have their first office visit after having initiated Valchlor.
  - Patients continuing treatment with Valchlor includes patients who are actively taking Valchlor on the day of enrollment.
  - Signed patient informed consent.

# Exclusion criteria:

None

# **VARIABLES**

The variables of interest for this study includes clinical characteristics, treatment patterns, clinical status, as assessed by the physician (including the methods used in practice to assess clinical status), MF-CTCL-related healthcare utilization, as assessed by the physician (hospitalizations and emergency room visits), AEs and


Doc No D-16.626


SAEs, patient-completed symptoms and QOL questionnaires.

Due to expected variability in practice patterns, no individual method of determining response is mandated, but assessments that do occur must be captured prospectively. Additionally, it is important to capture which methods were used pre-study, even where results may not be available, so that it is clear which assessments have a prior assessment that may have been considered in the physician's evaluation of response.

The specific outcomes and variables of interest for the study are:

Clinical characteristics.

Relevant medical history, including tumor-node-metastasis-blood (TNMB) classification.

Use of prior MF-CTCL treatments.

Treatment patterns, including prescribing information, for the treatment of MF-CTCL (including dosing regimens, titration schemes, duration of time from initiation to discontinuation of therapy, and drug holidays for Valchlor).

Clinical status, as assessed by the physician (i.e., complete response, partial response, stable disease, progressive disease, relapse).

Assessments (both whether or not the assessment was performed and the result of the assessment) used to define response, including, but not limited to:

- Composite Assessment of Index Lesion Severity (CAILS).
- Modified Severity Weighted Assessment Tool (mSWAT).
- Physician's Global Assessment.
- o Body Surface Area (BSA) of disease.

Healthcare utilization related to MF-CTCL during the study period, as assessed by physician:

- Number of MF-CTCL-related hospitalizations.
- Number of MF-CTCL-related emergency room visits.

AEs and SAEs (e.g., dermatitis) whether or not related to Valchlor.


MF-CTCL Doc No D-16.626


Patient-completed questionnaires:

- o Visual Analogue Scale (VAS) for pruritus (scale 0–10).
- o Skindex-29.
- o MF/SS CTCL.

# DATA SOURCES

Information will be collected per routine clinical practice. No specific clinical mandated assessments are to be performed as part of study participation. Patient-completed questionnaires, however, are a study requirement and will be collected at all clinic visits during the study observation period. These questionnaires will be administered on paper by study coordinators. Patient clinical data (non-patient-completed) will be collected from the patient's medical records at enrollment and throughout the study period. All data will be entered into electronic Case Report Forms (eCRFs) at the time of collection or on a quarterly basis by study coordinators. AEs and SAEs whether or not related to Valchlor will be entered into the eCRF at every visit and upon notification by the patient (e.g., reported via phone call).

For patients who do not have any visits, an affirmative response that the patient is still under care by the site will be requested quarterly, so that the absence of reported assessments can be interpreted the same as the actual absence of actual assessments.

**Pre-treatment** information will be collected at the time of enrollment using the following variables:

- Weight
- TNMB classification
- Use of Valchlor and other MF-CTCL treatments
- Assessments used to define response (whether or not the assessment was ever performed, and regardless of whether the assessment was used to assess response for a previously treated patient or whether the assessment was performed for a comparison with future evaluations of response, and the results of the most recent assessments), including, but not limited to:
  - o CAILS.
  - o mSWAT.
  - Physician's Global Assessment.
  - o BSA of disease.

In addition, the following information will be collected at the time

Doc No D-16.626


Version 3

# of enrollment:

Patient demographics.

Relevant medical history

MF-CTCL TNMB classification.

MF-CTCL histology.

Use of Valchlor and other MF-CTCL treatments (including start and stop dates for each medication, and reasons for starting and stopping medications).

Clinical status, as assessed by the physician (i.e., complete response, partial response, stable disease, progressive disease, relapse).

Assessments (both whether or not the assessment was performed and the result of the assessment) used to assess response, including, but not limited to:

- o CAILS.
- o mSWAT.
- o Physician's Global Assessment.
- o BSA of disease

All ongoing AEs and SAEs.

Patient-completed questionnaires:

- VAS for pruritus (scale 0–10).
- o Skindex-29.
- o MF/SS CTCL

The following information will be collected at all clinic visits occurring during the observation period:

MF-CTCL TNMB classification changes.

Changes in relevant medical history.

Use of Valchlor and other MF-CTCL treatments (including start and stop dates for each medication, and reasons for starting and stopping medications).

Healthcare utilization related to MF-CTCL since the last study visit, as assessed by physician:

o Number of MF-CTCL-related hospitalizations


MF-CTCL Doc No D-16.626


(including length of stay and primary admission and discharge diagnoses).

o Number of MF-CTCL-related emergency room visits.

Clinical status, as assessed by physician (i.e., complete response, partial response, stable disease, progressive disease, relapse).

Assessments (whether or not the assessment was performed and the result of the assessment) used to assess response, including, but not limited to:

- o CAILS.
- o mSWAT.
- o Physician's Global Assessment.
- BSA of disease.

All AEs and SAEs (e.g., dermatitis) whether or not related to Valchlor, including reports of secondary exposures since last visit (while on Valchlor only).

Patient-completed questionnaires:

- VAS for pruritus (scale 0–10).
- o Skindex-29.
- o MF/SS-CTCL.

Patients who enrolled under the original protocol and are still ongoing in the study will be contacted and informed consent will be obtained for the Amendment 1 protocol. Patients prospective data will be collected up to a total of 24 months from the original enrollment date.

### STUDY SIZE

This study will enroll approximately 300 patients diagnosed with MF-CTCL who are being treated with Valchlor.

A sample size of 270 evaluable patients is needed to estimate the percentage of patients with clinical status and the rate of hospitalizations, both with a margin of error of 6 percentage points. Assuming that up to 10% of patients may be non-evaluable due to incomplete follow-up, the sample size target for enrollment should be 300. It is projected that approximately 200 evaluable patients currently enrolled will be re-consented and newly enrolled will be consented under Amendment 1 for a 2-year follow-up. The margin of error for 200 evaluable patients will be 7%.

Additionally, it is important to be able to estimate these same

Doc No D-16.626


| | percentages with a margin of error of 10 percentage points or less for key subgroups representing a third or more of the patient population (e.g., patients newly initiating Valchlor). A total of 100 patients are required to achieve a margin of error of 10 percentage points, so that a total enrollment of 300 patients is needed. |
|---|---|
| DATA<br>ANALYSIS | Demographics and clinical characteristics will be summarized for all patients enrolled as well as grouped separately for patients continuing treatment with Valchlor versus patients who are newly initiating Valchlor. Use of prior treatments and past methods of assessing response will similarly be analyzed separately for the two groups. Treatments individually and in combination will be reported in percentage terms, by visit, stratified by newly initiating patients and continuing patients to identify treatment patterns. |
| | Analyses of response, based on a particular measure of response, will be limited to patients for whom that measure was reported. Therefore, patients with reported data will be summarized also for patients without any reported data with respect to demographics and pre-treatment clinical status to identify potential biases. Rates of on-study hospitalization and emergency room visits will be computed as the utilization counts divided by on-study days. The summary of response rates will be tabulated and the definition of response will be detailed in the Statistical Analysis Plan. |
| | The frequency and percentage of patients experiencing any AEs or SAEs will be summarized by system organ class and preferred MedDRA terminology. SAEs requiring hospitalizations and fatal SAEs will be displayed in patient listings. |
| | At each visit performed during the observation period (1 <sup>st</sup> , 2 <sup>nd</sup> , etc.), the VAS for pruritus, the three scales of the Skindex-29 and the MF/SS-CTCL questionnaires will be computed for patients who are and are not responders. These descriptive cross-sectional comparisons are intended to assess burden of disease in a Valchlor-treated cohort over time. |
| MILESTONES | First patient, first visit: Q4 2014 |
| | Last patient, first visit: Q3 2017 |
| | Last patient, last visit: Q3 2019 |

Epidemiology and Observational Studies AC-079A501 Version 3


| DATA | Actelion Pharmaceuticals US, Inc. |
|---|---|
| OWNERSHIP | |
| STUDY | The Scientific Committee will consist of 4–6 key opinion leaders in |
| COMMITTEE(S) | the field of MF-CTCL who will provide scientific input on the |
| | MF-CTCL Study protocol and review study data. |


Version 3

# 13 December 2016, page 17/43

# **PROTOCOL**

# 1 AMENDMENTS AND UPDATES (PROTOCOL HISTORY)

The protocol version 2, dated 12 November 2014, Appendix A, Appendix B and section 5.7.6 for the Skindex-29 Questionnaire were updated. As these were administrative changes, no amendment was required; only a new protocol version number was issued. The protocol Amendment 1 will originate version 3 to extend ongoing patients and newly enrolled patients for a total of 24 months from consent date. An additional new quality of life assessment has been added.

# 2 STUDY MILESTONES

This study will be conducted according to the following schedule:

First patient, first visit: Q4 2014 Last patient, first visit: Q3 2017 Last patient, last visit: Q3 2019

# 3 RATIONALE AND BACKGROUND

# **Background**

Mycosis fungoides cutaneous T-cell lymphoma (MF-CTCL) can present as patches, plaques, or tumors on the skin, often in areas of the body that are not usually exposed to the sun [Lymphoma.org 2011]. While MF-CTCL is rare, it is the most common type of cutaneous T-cell lymphoma (CTCL), accounting for 50–70% of all CTCLs [Imam 2013]. It is estimated that approximately 16,000 to 20,000 people in the US have the disease and that the 5-year incidence of MF-CTCL for all stages was 0.56 per 100,000 person-years between 2005–2009 [Korgavkar 2013, Leukemia & Lymphoma Society 2011]. The prevalence and incidence of MF-CTCL are likely to be under-reported due to nomenclature variances and because the symptoms and skin biopsy findings can appear similar to other types of skin conditions [Lymphoma.org 2011, Criscione 2007]. Patients frequently present with early stage disease typically associated with a favorable prognosis and survival of 10–35 years, but over 25% progress to advanced disease with a median survival of less than 4 years and just 13 months in those with nodal involvement [Scarisbrick 2014]. The most important clinical predictive factors for survival include patient age, T classification, and the presence of extracutaneous disease [Kim 2003a].

Although there is currently no cure for the disease, patients diagnosed at early stages of MF-CTCL (Stages IA, IB, or IIA) and receiving treatment for the disease have a median survival of 35.5, 21.5, and 15.8 years, respectively [Agar 2010]. Topical mechlorethamine hydrochloride (MCH or nitrogen mustard) has been used to treat


MF-CTCL Doc No D-16.626


MF-CTCL since the 1950s [Lessin 2013]. The National Comprehensive Cancer Network [NCCN] Guidelines list topical MCH as a primary skin-directed treatment option for patients with MF-CTCL with limited/localized skin involvement or for generalized skin involvement [NCCN 2014]. Topical MCH has been available in aqueous and petrolatum-based forms. However, both forms have disadvantages that limit patient acceptance [Kim 2003b, Ramsay 1995].

Valchlor, approved by the FDA in August 2013 for Stage IA and IB MF-CTCL, is a fast-drying, greaseless gel formulation that has been shown to be effective and safe in a clinical trial [Lessin 2013]. Two hundred sixty (260) patients in the Valchlor clinical trial (Study 201) received MF-CTCL specific treatment up to 12 months [Lessin 2013]. In the open-label, single group extension trial, 98 patients who completed Study 201 without a complete response received treatment with a formulation identical to Valchlor but containing MCH HCl 0.04% for 7 months. Currently, Valchlor is the only FDA-approved formulation of topical MCH, and one of two FDA-approved topical treatments for MF-CTCL [Kim 2014]. The results of the randomized, controlled, multi-center trial confirmed the non-inferiority of Valchlor in the treatment of MF-CTCL when compared to ointment-based MCH.

### Rationale

Prospective data on Valchlor are currently only available from the pivotal, randomized, controlled clinical trial with strict inclusion and exclusion criteria. Understanding real-world patient safety and tolerability, as well as compliance and discontinuation rates, will assist with the future management of Valchlor-treated MF-CTCL patients. This study will build and extend on the data from the Valchlor clinical development program, increase the understanding of the use of Valchlor in patients with MF-CTCL and, while limited to patients treated with Valchlor, will represent the largest prospective study with any given MF-CTCL treatment.

This large, non-interventional study will provide information on the use of Valchlor in a 'real-world' clinical practice setting. This study will increase understanding of the management and outcomes of Valchlor-treated MF-CTCL patients by observing clinical characteristics, treatment patterns, outcomes (e.g., clinical status and healthcare utilization [MF-CTCL-related hospitalizations and emergency room visits]), and adverse events (AEs). Additionally, a better understanding of the disease burden of MF-CTCL will be gained by collecting patient-completed symptoms and quality of life (QOL) questionnaires.

# 4 RESEARCH QUESTION AND OBJECTIVES

The objectives of the MF-CTCL prospective cohort study are:

Epidemiology and Observational Studies AC-079A501 Version 3 13 December 2016, page 19/43


- To describe clinical characteristics of patients treated with Valchlor at enrollment and during the study observation period.
- To describe treatment and response assessment patterns of patients with MF-CTCL treated with Valchlor at enrollment and during the study observation period.
- To assess outcomes (e.g., clinical status and rates of healthcare utilization [MF-CTCL-related hospitalizations and emergency room visits]) in patients with MF-CTCL treated with Valchlor during the study observation period.
- To collect and describe the incidence of AEs/SAEs in patients with MF-CTCL treated with Valchlor:
  - To estimate the incidence of dermatitis in patients using Valchlor during the study observation period.
  - o To describe the management of dermatitis in patients using Valchlor at enrollment and during the study observation period.
- To collect patient-completed symptoms and QOL questionnaires.

# 5 RESEARCH METHODS

# 5.1 Study design

This is a multi-center, prospective, observational study of MF-CTCL patients who have newly initiated Valchlor or who are continuing treatment with Valchlor.

Patients will be followed by their physician according to routine clinical practice. With the exception of protocol-required patient-completed questionnaires, there are no specific or mandated clinical assessments to be performed, and patients will not receive experimental intervention or treatment as a consequence of their participation in this study. The study protocol will not mandate any specific schedule of visits. Patients will undergo clinical assessments and receive standard medical care as determined by the patient's physician in a real-world setting.

Patients will be followed prospectively for a maximum of 2 years from the date of signed informed consent until end of study (EOS), which includes withdrawal of consent, loss to follow-up, death, or study completion. Continuation in the study is not continuent on continuation of Valchlor.

The study will end after all enrolled patients have been followed for 2 years, or discontinued from the study for any reason.

# 5.2 Population (setting and study population)

This study will enroll approximately 300 MF-CTCL patients being treated (newly initiated or continuing treatment) with Valchlor [see Section 5.2.1 for details] from up to 50 participating centers/clinics in university-affiliated or community hospitals.


Epidemiology and Observational Studies AC-079A501 Version 3 13 December 2016, page 20/43

Patients considered 'being treated with Valchlor' is comprised of two distinct groups: 1) Patients newly initiating Valchlor. These are patients who are enrolled at their first office visit after having initiated Valchlor; 2) Patients continuing treatment with Valchlor. Patients must be actively taking Valchlor on the day of enrollment.

All consecutive MF-CTCL patients being treated with Valchlor [see Section 5.2.1 for details] seen at the participating centers are eligible for enrollment in the study, regardless of other MF-CTCL therapies received before or at the time of enrollment.

### 5.2.1 Inclusion criteria

- All adult patients (≥ 18 years of age) diagnosed with MF-CTCL and being treated with Valchlor. This includes patients newly initiating Valchlor OR patients continuing treatment with Valchlor:
  - o Patients newly initiating Valchlor are patients who have their first office visit after having initiated Valchlor.
  - o Patients continuing treatment with Valchlor includes patients who are actively taking Valchlor on the day of enrollment.
- Signed patient informed consent.

# 5.2.2 Exclusion criteria

None.

### 5.3 Variables

The variables of interest for this study includes clinical characteristics at enrollment and during the study observation period, treatment patterns, clinical status, as assessed by the physician (including the methods used in practice to assess clinical status), MF-CTCL-related healthcare utilization, as assessed by the physician (hospitalizations and emergency room visits), AEs and SAEs, patient-completed symptoms and QOL questionnaires.

Data elements to be collected from the patient's medical record at study enrollment and at post-enrollment follow-up visits are shown in Table 1. Additionally, pre-treatment data collection using specific variables will be performed at enrollment. These variables include weight, tumor-node-metastasis-blood (TNMB) classification, use of Valchlor and other MF-CTCL treatments, and clinical status assessments. Drug holidays (temporary discontinuation) from Valchlor will be captured on the electronic Case Report Form (eCRF) by recording start and stop dates of all MF-CTCL treatments. Patient-completed questionnaires will be administered to patients who can read and understand English or Spanish and are able to self-complete the questionnaires based on the investigator's assessment. Patients who are unable to read and understand English or Spanish will not be asked to complete the questionnaires and will be excluded from the study.

Epidemiology and Observational Studies AC-079A501 Version 3

MF-CTCL


Table 1 eCRF Data Collection

| Variables | Enrollment visit | Post-enrollment follow-up visits |
|---|---|---|
| Informed Consent | X | $X^1$ |
| Demographics | | |
| Age, gender, race/ethnicity, height | X | |
| Weight* | X | |
| Relevant Medical History | | |
| Age at diagnosis of MF-CTCL | X | |
| Date of MF-CTCL diagnosis | X | |
| Method of diagnosis | X | |
| MF-CTCL TNMB classification* | X | |
| MF-CTCL TNMB classification change | | X |
| MF-CTCL histology | X | |
| Malignancies and secondary malignancies | X | |
| Non-melanoma skin cancers | X | |
| Prior viral infections | X | |
| Atopic disorders | X | |
| Psoriasis | X | |
| Urticaria | X | |
| Mental disorders | X | |
| Family medical history | X | |
| Other relevant medical history | X | |
| Changes in medical history | | X |
| Targeted MF-CTCL Treatments (Medication Use and Dosing)* $^{\dagger}$ | _ | |
| Valchlor | X | X |
| Other MF-CTCL treatments | X | X |

# MF-CTCL Epidemiology and Observational Studies AC-079A501 Version 3


| Variables | Enrollment visit | Post-enrollment follow-up visits |
|---|---|---|
| Healthcare utilization related to MF-CTCL (as assessed by physician) | | |
| Hospital admissions <sup>‡</sup> | | X |
| Emergency room visits | | X |
| Clinical Status (as assessed by physician) | X | X |
| Clinical Status Assessments* | | |
| Composite Assessment of Index Lesion Severity | X | X |
| Modified Severity Weighted Assessment Tool | X | X |
| Physician's Global Assessment | X | X |
| Body Surface Area of disease | X | X |
| Patient-Completed Questionnaires <sup>§</sup> | | |
| Visual Analogue Scale for pruritus | X | X |
| Skindex-29 | X | X |
| Mycosis fungoides / Sézary syndrome-type cutaneous T-cell lymphoma | X | X |
| Safety Measures** | | |
| AEs and SAEs | $\mathbf{X}^{+}$ | X |
| Reports of secondary exposures | | $\mathbf{X}^{^{\wedge}}$ |

<sup>\*</sup>Included in pre-treatment data collection, which is performed at enrollment. All data must be completed as available

<sup>&</sup>lt;sup>†</sup>Includes collection of start and stop dates for each medication, including reasons for starting and stopping medications. Start and stop dates are also collected for Valchlor, including short gaps in treatment, such as drug holidays.

<sup>&</sup>lt;sup>‡</sup>For each hospital admission, length of stay and primary admission and discharge diagnoses will be collected.

<sup>§</sup>To be completed by patients who can read and understand English and are able to self-complete the questionnaires based on the investigator's assessment. Patients who are unable to self-complete the questionnaires will not be excluded from the study.

<sup>\*\*</sup>Safety measures, which include AEs and SAEs, will be collected from the informed consent date and prospectively at every visit during the study and up to 30-days post-discontinuation of Valchlor during the study. Ongoing AE and SAE data will be collected through the end of study, regardless of Valchlor use.

MF-CTCL Epidemiology and Observational Studies AC-079A501 Version 3


Doc No D-16.626


New AEs and SAEs that occur more than 30 days after discontinuation of Valchlor will be reported to Actelion US Drug Safety if investigator feels there is a possible causal relationship with Valchlor. Investigators are also expected to assess patients for AEs and SAEs and follow the appropriate reporting procedures per Section 7.

<sup>†</sup>All ongoing AEs and SAEs for patients being treated [see Section 5.2.1 for definition of "being treated"] with Valchlor.

All reports of secondary exposures, as available, will be counted on the eCRFs. Additional information regarding secondary exposures will be forwarded directly to Actelion US Drug Safety via the Secondary Exposure Form. Refer to Section 7.1.1 for definition of secondary exposure.

AE = adverse event; eCRF = electronic Case Report Form; MF-CTCL = mycosis fungoides cutaneous T-cell lymphoma; SAE = serious adverse events; TNMB = tumor-node-metastasis-blood.

<sup>1</sup>Re-consent at the first follow up visit for subjects who are currently active in the study prior to Amendment 1.

### **5.3.1** Outcome definition and measures

The clinical outcomes and variables of interest for this study are clinical characteristics, treatment patterns, clinical status, as assessed by the physician (and the methods used in practice to assess clinical status), MF-CTCL-related healthcare utilization, as assessed by the physician (hospitalizations and emergency room visits), AEs and SAEs (e.g., dermatitis), and patient-completed symptoms and QOL questionnaires. Due to expected variability in practice patterns, no individual method of determining response, either at follow-up or in tandem with a prior assessment, is mandated and a subjective categorical assessment of response will be included in addition to quantitative measures of response, but assessments that do occur must be captured prospectively. Additionally, it is important to capture which methods were used pre-study, even where results may not be available, so that it is clear which assessments have a prior assessment that may have been considered in the physician's evaluation of response.

For patients who do not have any assessments, an affirmative response that the patient is still under care by the site will be requested quarterly so that the absence of reported assessments can be interpreted the same as the absence of actual assessments.

The following specific outcomes and variables of interest will be evaluated:

Clinical characteristics at enrollment and during study observation period.

Relevant medical history, including TNMB classification.

Use of prior MF-CTCL treatments.

Treatment patterns, including prescribing information, for the treatment of MF-CTCL (including dosing regimens, titration schemes, duration of time from initiation to discontinuation of therapy, and drug holidays for Valchlor).

Clinical status, as assessed by the physician (i.e., complete response, partial response,

Epidemiology and Observational Studies AC-079A501 Version 3


stable disease, progressive disease, relapse).

Assessments (both whether or not the assessment was performed and the result of the assessment) used to define response, including, but not limited to:

- Composite Assessment of Index Lesion Severity.
- o Modified Severity Weighted Assessment Tool.
- o Physician's Global Assessment.
- o Body Surface Area of disease.

Healthcare utilization related to MF-CTCL during the study period, as assessed by physician:

- o Number of MF-CTCL-related hospitalizations.
- o Number of MF-CTCL-related emergency room visits.

AEs and SAEs (e.g., dermatitis) whether or not related to Valchlor.

Patient-completed questionnaires:

- Visual Analogue Scale for pruritus (scale 0–10).
- o Skindex-29.
- Mycosis fungoides / Sézary syndrome-type cutaneous T-cell lymphoma (MF/SS-CTCL).

# **5.3.2** Exposure definition and measures

Start of observation is defined as date of signed informed consent.

End of observation is defined as EOS, including death, withdrawal of consent, loss to follow-up, or study completion, whichever occurs first.

Total exposure time is defined as the date of first Valchlor exposure to the date of last Valchlor exposure.

Total on-study Valchlor exposure time is defined as the first day of Valchlor use to last day of Valchlor use during the observation period. If the patient was using Valchlor at end of observation, the last on-study day of Valchlor use is equal to the end date of observation period. Drug holidays are excluded from the sum of exposure time.

# **5.3.3** Covariate definition and measures

The following covariates will be considered for analyses as well as for exploring their relationship to safety-related (e.g., dermatitis) outcomes:

Age at enrollment, gender, race/ethnicity.

MF-CTCL medical history:

o Time since diagnosis and TNMB classification.


Version 3

Medical history of previous and ongoing clinically significant underlying diseases and comorbid conditions.

Prior exposure to Valchlor and other MF-CTCL specific therapies.

### 5.4 Data sources

Data elements to be collected include the following: patient demographics, personal and family medical history, including MF-CTCL diagnosis date and etiology, current and historical MF-CTCL treatments, clinical status (as assessed by the physician), and which assessments were used to define response, MF-CTCL-related healthcare utilization (as assessed by the physician), AEs and SAEs whether or not related to Valchlor, deaths, patient-completed symptoms and QOL questionnaires. Table 1 provides an overview of the variables collected at enrollment and during the observation period [see Section 5.3.2 for definition]. For patients who do not have any visits, an affirmative response that the patient is still under care by the site will be requested quarterly, so that the absence of reported assessments can be interpreted the same as the absence of actual assessments.

Since this is a real-world, observational study, there are a number of sources of bias that could potentially affect any conclusions that may be drawn. The methods used to minimize these sources of bias in this study are detailed below [see Section 5.9].

Therapies specific to MF-CTCL during the course of this study are under the direction of the participating physician and not the study protocol. As this study collects data on both incident patients and prevalent patients, it is necessary to include the date of diagnosis in the data collection forms, in order to minimize potential survivor bias effect.

# 5.5 Study size

This study will have an approximate enrollment of 300 patients diagnosed with MF-CTCL who are being treated with Valchlor (newly initiated or continuing treatment).

A sample size of 270 evaluable patients is needed to estimate the percentage of patients with clinical status and the percentage of patients with hospitalizations, both with a margin of error of 6 percentage points. Assuming that up to 10% of patients may be non-evaluable due to incomplete follow-up, the sample size target for enrollment should be 300.

It is projected that approximately 200 evaluable patients will be re-consented under Amendment 1. The margin of error for 200 evaluable patients will be 7%.

Additionally, it is important to be able to estimate these same percentages with a margin of error of 10 percentage points or less for key subgroups representing a third or more of the patient population (e.g., patients newly initiating Valchlor). A total of 100 patients are required to achieve a margin of error of 10 percentage points per subgroup, so that a total enrollment of 300 patients is needed.


Doc No D-16.626

# 5.6 Data management


# 5.6.1 Data collection

Version 3

Informed consent must be obtained prior to enrollment and data collection.

Re-consent must be obtained for patients that were enrolled in the study prior to Amendment 1 and still ongoing to complete 24 months of data collection from the enrollment date. Instead of the 12 months initially planned.

This study will collect data on MF-CTCL patients being treated with Valchlor [see Section 5.2.1 for inclusion criterial under routine clinical care. This will include both data collected from assessments that are routinely performed for MF-CTCL patients being treated with Valchlor in clinical practice, and additional data from further assessments that may be performed.

No specific clinically mandated assessments are to be performed as part of study participation. Patient-completed questionnaires, however, are a study requirement and will be collected at all clinic visits during the study observation period. These questionnaires will be administered on paper by study coordinators. Patient clinical data (non-patient-completed) will be collected from the patient's medical records at enrollment and throughout the study period. All data will be entered into an eCRF at the time of collection or on a quarterly basis by study coordinators. AEs, reports of secondary exposure, and SAEs whether or not related to Valchlor will be entered into the eCRF at every visit and upon notification by the patient (e.g., reported via phone call).

A secure, Internet-based electronic data collection (EDC) system will be used for data entry and hosting. An audit trail will be maintained by the EDC system for all data entries and changes, indicating what entries/changes have been made, who made them, and when. Data will be encrypted when transferred over the Internet and will be stored in a secure database protected from unauthorized access.

All data collected will be de-identified before transmission to the central study coordinating center. Patient names will not be collected. Other patient identifiers will be collected in order to allow identification of study patients when SAEs are received by US Drug Safety outside of the study [see Section 7.4].

All SAE data entered into the Adverse Event (AE)/Adverse Drug Reaction (ADR) Form and all reports of secondary exposure will be transferred electronically and/or by fax by the physician to Actelion US Drug Safety to be processed in the Actelion Drug Safety Database. In addition, all AE data, reports of secondary exposure, and SAE data will be entered into the study eCRF.


# 5.7 Data analysis


# **Analysis sets and groups**

Demographics and clinical characteristics will be summarized for all enrolled patients and also grouped separately for patients continuing treatment with Valchlor versus patients who are newly initiating Valchlor. Use of prior treatments and past methods of assessing response will be similarly analyzed separately for the two groups. The methods used for assessment of response (i.e., assessed with that method versus not assessed with that method, either at follow-up alone or in tandem with a prior assessment) will be reported as cumulative percentages over time and also as a percentage of first visits, second visits, etc. To minimize the potential impact of missing data, analyses will focus on variables that are available for all patients, such as whether a particular type of assessment occurred, rather than focusing on the results of a particular assessment. Analyses of response, based on a particular measure of response, will be limited to patients for whom that measure was reported. Therefore, patients with reported data will be compared to patients without any reported data with respect to demographics and pre-treatment clinical status to identify potential biases. The summary of response rates will be tabulated and the definition of response will be detailed in the Statistical Analysis Plan.

#### 5.7.2 Clinical characteristics

Analyses of prior treatment, assessments, and relevant medical history will be summarized for all patients enrolled and also grouped separately for patients newly initiating Valchlor versus patients continuing on Valchlor. Percentages will generally be computed as a function of non-missing data; however, if a large amount of data are missing for some historical data, a comparison of patients with missing and non-missing data may be necessary to ensure generalizability based on non-missing data alone.

# 5.7.3 Treatment and assessment patterns

Because relatively little prospectively collected data is available on MF-CTCL treatment patterns, preliminary analysis will make use of patient listings to develop categories of treatment patterns. Categories will be developed without cross-referencing outcomes data to minimize bias (i.e., the focus will be the presence of specific assessments, not the test value associated with the assessment). Treatments individually and in combination will be reported in percentage terms, by visit, stratified by newly initiating patients and continuing patients to identify treatment patterns.

Duration of time from first post-initiation of Valchlor office visit to discontinuation of therapy will be assessed using Kaplan-Meier estimates of freedom from discontinuation. If short-term gaps in therapy are common, sensitivity analyses may be conducted in which these gaps do or do not count as treatment discontinuations, depending on the lengths of the gaps. These analyses will focus only on newly initiated patients.


Version 3


# 5.7.4 Clinical outcomes

The main clinical outcomes that will be analyzed are clinical response, as assessed by the physician, and MF-CTCL-related healthcare utilization, as assessed by the physician (e.g., hospitalizations and emergency room visits). Rates of on-study hospitalization and emergency room visits will be computed as the ratio of utilization counts divided by on-study days. Hospitalization-free survival will be computed using Kaplan-Meier estimates.

Because a wide variation in assessments of clinical response is expected, the clinician's subjective evaluation of response will be summarized in addition to reporting the proportion of responses among patients for whom specific tests were performed. The subjective response will be cross-classified by which assessments were used. The summary of response data is primarily a descriptive analysis to better understand how and when physicians define response, and it does not represent an estimate of the efficacy of any MF-CTCL treatment.

### 5.7.5 Adverse events

The frequency and percentage of patients experiencing any on-study AEs, SAEs, or death will be summarized by system organ class and preferred MedDRA terminology. Additional detail for AEs of special interest (e.g., dermatitis) will be summarized separately. SAEs will be displayed in patient listings, both including and excluding events that were not concurrent with Valchlor exposure. The definition of an on-study event is one that occurs on the day of enrollment or later, but before the date of study discontinuation or completion.

# **5.7.6** Patient-completed questionnaires

The Skindex-29 is a questionnaire that results in three scales: emotions, symptoms, and functioning [Chren 1996, Chren 1997a, Chren 1997b, Chren 2001]. Appendix A shows the items in the Skindex-29 questionnaire and Appendix B describes the scoring of individual items to the 3 scales. To compute the scale, each item is first transformed to a linear 0–100 scale where responses of "Never", "Rarely", "Sometimes", "Often", and "All the time" are converted to values of 0, 25, 50, 75, and 100, respectively. Next, the mean of the non-missing items for each scale is computed to derive a scale score. Although missing data for individual items is allowed, no scale score will be computed if more than quarter of the items in the scale are missing.

The VAS for pruritus is a single value [Reich 2012] and is shown in Appendix C.

The MF/SS-CTCL questionnaire contains 12 questions [PatientsLikeMe 2016] and is shown in Appendix D.

At each study visit (1<sup>st</sup>, 2<sup>nd</sup>, etc.), the VAS for pruritus, the three scales of the Skindex-29 and the MF/SS-CTCL will be computed for patients who are and are not responders,


Version 3

based on clinician assessment, at the time of that visit. These descriptive cross-sectional comparisons are intended to assess burden of disease in a Valchlor-treated cohort over time. The data related to all three questionnaires (VAS, Skindex-29, MF/SS-CTCL) will be collected on the QOL questionnaires.

# 5.8 Quality control

The use of the EDC system will allow for on-line data quality checks upon data entry. The EDC system will have pre-programmed automatic edit checks for data inconsistencies at the time of data entry, and resulting queries will be addressed by the site.

Site visits may be conducted by Actelion or by an authorized Actelion representative to inspect study data, patient medical records, and eCRFs.

No source data verification is mandated. However, the data will be reviewed on an ongoing basis for implausible data points, missing data points, assessments not conducted, and/or incomplete information. This review may result in queries to the sites. Centralized remote monitoring of patient data will be performed via the EDC tool. This approach will allow proactive monitoring and querying of data on an ongoing and regular basis with concentrated efforts on key data points (e.g., hospitalization, death, Valchlor interruption and discontinuation, AEs and SAEs, and secondary exposures) to encourage low rates of missing information. Communication with investigators and study coordinators will emphasize the importance of data entry completion. Analytical methods described in Section 5.7 will be applied to assess the extent of the missing data and the impact on inferential estimates.

# 5.9 Discussion of the study methods (including limitations)

This study is an observational, prospective study examining MF-CTCL patients being treated with Valchlor in a real-world clinical setting. Valchlor treatment will be based on prescriber decision and will not be influenced by participation in this study. The patients will be followed by their physician according to routine clinical practice. The study protocol does not mandate any treatment, procedures or visits. Patient-completed questionnaires, however, are a study requirement and will be administered at all study visits for patients who can read and understand English, and are physically and mentally able to complete the questionnaires based on the investigator's assessment.

Any interpretation of observational study results should consider limitations to observational real-world study designs, including potential sources of selection or information biases, and confounding factors.

To minimize selection bias, participating centers will offer enrollment in the study to all consecutive MF-CTCL patients currently treated with Valchlor [see Section 5.2.1 for inclusion criteria], regardless of other MF-CTCL specific therapy received before or at


Version 3

the time of enrollment, or during the study. This study collects data on all users of Valchlor. At enrollment, a review of existing medical records will be performed to collect information as described per Table 1 (enrollment visit). Thereafter, all data will be collected during the observation period.

Patients who are enrolled under the original protocol prior to protocol Amendment 1 and are still ongoing in the study will be re-consented under Amendment 1 and will continue to follow the schedule of Table 1 eCRF Data Collection specified in this protocol up to end of study (Month 24). Patients who enrolled and have completed 1 year of the study under the original protocol will not be offered to continue in the study and thus not re-consented under Amendment 1.

To minimize the number of patients lost to follow-up, there will be regular contact with patients by the site, including 3 attempts to contact a patient before she/he is considered lost to follow-up.

# 6 PROTECTION OF HUMAN SUBJECTS AND ETHICAL APPROVAL

# 6.1 Institutional Review Board/Independent Ethics Committee approval

Depending on local regulations and the physician's institutional policies, and in compliance with local law, the physician may have to submit the study protocol, the form for the Patient Informed Consent, and other relevant information to an Institutional Review Board (IRB) / Independent Ethics Committee (IEC), local health authorities, data protection agency or others. Approval from the IRB/IEC must be obtained before going through a consent procedure with the patient and before entering data into the database. IRB/IEC information/approval must be documented in a letter to the physician, clearly identifying the study, the documents reviewed, and the date of approval.

# 6.2 Patient informed consent

The participating physician commits to obtaining approval for the Patient Informed Consent Form from his/her respective Research Ethics Board, if required by applicable site policies, national privacy regulations and other state and local laws relating to medical information, prior to commencement of the project. Moreover, if required, the participating physician will obtain a signed Patient Informed Consent Form from each patient (or legal guardian) whose data will be included in the project.

# **6.3** Patient confidentiality

By signing the protocol, the participating physician commits to complying with all related applicable local laws and regulations, including but not limited to the regulations in 45 CFR parts 160 and 164 (protected health information), such regulations also known as the "HIPAA Privacy Regulations".

Doc No D-16.626

Version 3


#### MANAGEMENT AND REPORTING OF ADVERSE EVENTS 7

With reference to collecting, processing and expediting of AE reports, Actelion as the sponsor of this prospective non-interventional study complies with international and national pharmacovigilance regulations.

# 7.1 Definitions

# 7.1.1 Adverse event or adverse experience

Any untoward medical occurrence in a patient administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.

### AEs include:

Recurrence or worsening of a pre-existing disease.

Increase in frequency or intensity of symptoms of a pre-existing disease or medical condition.

Continuous persistent disease or symptoms present at initiation of treatment or enrollment, which occurs first, that worsen following the start of the study.

Lack of efficacy in the acute treatment of a life-threatening disease Abnormal assessments, e.g., ECG, vital signs, or physical examination findings, if they represent a clinically significant finding that was not present at initiation of treatment or enrollment, which occurs first, or worsened during the course of the study or led to dose reduction, interruption or permanent discontinuation of Valchlor.

Laboratory test abnormalities if they represent a clinically significant finding, symptomatic or not, which were not present at initiation of treatment or enrollment, which occurs first, or worsened during the course of the study or led to dose reduction, interruption or permanent discontinuation of Valchlor.

In addition to AEs, exposure during pregnancy or lactation, product complaints, medication errors, overdose, misuse, abuse, occupational exposure and transmission of an infectious agent via Valchlor and the identification of a potential counterfeit medicinal product needs to be reported.

Reports of off-label use without an associated AE collected within non-interventional studies shall be included in final study reports.

Reports of inadvertent secondary exposure to the skin, mucous membranes, and eyes of individuals other than the patient being treated (e.g., patient's caregiver or family member).

Epidemiology and Observational Studies AC-079A501 Version 3 13 December 2016, page 32/43


AEs do not include:

Medical procedures such as surgery, endoscopy, tooth extraction. However, the event that led to the intervention is considered an AE.

Situations in which no undesirable change occurred, such as hospitalization for cosmetic surgery or for social reasons.

### 7.1.2 Serious adverse events

An SAE is defined by the International Conference on Harmonisation guidelines as any AE fulfilling at least one of the following criteria:

Fatal.

Life-threatening: refers to an event in which the subject was at risk of death at the time of the event. It does not refer to an event that hypothetically might have caused death had it been more severe.

Requiring inpatient hospitalization, or prolongation of existing hospitalization.

Resulting in persistent or significant disability or incapacity.

Congenital anomaly or birth defect.

Medically significant: refers to important medical events that may not immediately result in death, be life-threatening, or require hospitalization but may be considered to be SAEs when, based upon appropriate medical judgment, they may jeopardize the subject, and may require medical or surgical intervention to prevent one of the outcomes listed in the definitions above

The following reasons for **hospitalizations** are exempted from being reported:

Hospitalizations for cosmetic elective surgery, or social and/or convenience reasons.

Hospitalization for pre-planned (prior to enrollment) standard monitoring of a pre-existing disease (present at enrollment) or medical condition that did not worsen, e.g., hospitalization for coronary angiography in a patient with stable angina pectoris.

Hospitalizations for elective treatment of a pre-existing disease (present at enrollment) or medical condition that did not worsen, e.g., elective hip replacement for arthritis.

New AEs and SAEs that occur > 30 days after the discontinuation of Valchlor unless there is a reasonable possibility of causal relationship to Valchlor.

However, complications that occur during such hospitalizations are AEs or SAEs (for example, if a complication prolongs hospitalization) and must be reported as described below.

Epidemiology and Observational Studies AC-079A501 Version 3 13 December 2016, page 33/43


# 7.1.3 Relationship to the use of Valchlor

Each AE must be assessed by the investigator as to whether or not there is a reasonable possibility of causal relationship to Valchlor, and reported as either related or unrelated. The determination of the likelihood that Valchlor caused the AE will be provided by an investigator who is a qualified physician.

# Related to Valchlor

This category applies to any AE (whether serious or not) that appears to have a reasonable possibility of causal relationship to the use of Valchlor (i.e., a relationship cannot be ruled out). Guidelines to determine whether an event might be considered related include (but are not limited to) the following:

There is temporal relationship between the occurrence of the event and the administration of Valchlor

The event abated (diminished) or disappeared when treatment with Valchlor was down-titrated, interrupted, or discontinued.

The event recurred when treatment was re-introduced.

### Unrelated to Valchlor

This category applies to any AE (whether serious or not) that does not appear to have a reasonable relationship to the use of Valchlor (see above guidelines). Environmental factors such as clinical state and other treatments could equally have caused the event.

# 7.2 Secondary exposures, AE and SAE reporting to Actelion US Drug Safety

All reports of secondary exposures and all AEs will be recorded on the eCRFs and captured in the EDC clinical database. The AE data will be forwarded to Actelion US Drug Safety at predetermined intervals.

All SAEs (including secondary exposures) which occur after initiation of Valchlor treatment until 30 days after Valchlor discontinuation must be collected, recorded and reported during the study. New AEs and SAEs that occur more than 30 days after the discontinuation of Valchlor will be reported to Actelion US Drug Safety if the investigator assesses that there is a possible causal relationship with Valchlor. The minimum information required for collecting and forwarding an SAE to Actelion US Drug Safety is the product name, patient identifier, reporter contact information, and the identified SAE. All SAEs must be recorded on an AE/ADR Form. Cases of secondary exposure must recorded on the Secondary Exposure Form and submitted directly to Actelion US Drug Safety. The AE/ADR Form will be pre-populated with the information already entered in the eCRF, and it is the physician's responsibility to complete, print, and sign the form and forward to Actelion US Drug Safety directly, within 1 working day

Epidemiology and Observational Studies AC-079A501 Version 3


of the investigator's first knowledge of the event, by fax or using the drug safety email address:


Doc No D-16.626

FAX: (866) 227-5886 Actelion US Drug Safety: drugsafetyUS@actelion.com

Actelion US Drug Safety will acknowledge the receipt of the AE/ADR form and provide a Manufacturer's Control Number (MCN – a unique number assigned by Drug Safety's database to the case) to the investigator and the Actelion Operations (Clinical Study Leader) within 48 hours. If no acknowledgement is received from Actelion US Drug Safety, the investigator must follow up immediately (or within 1 working day) with a phone call or email to Actelion US Drug Safety to ensure the AE/ADR Form has been received.

# 7.2.1 Follow-up of SAEs

Actelion US Drug safety will evaluate and process all safety reports received. If follow-up information is required, Actelion US Drug Safety will send a Data Clarification Form (DCF) directly to the investigator.

Follow-up information about a previously reported SAE must be reported directly to Actelion US Drug Safety via the AE/ADR Form within 1 working day of the investigator's first knowledge of the event.

If the subject is hospitalized in a hospital other than the study site, it is the investigator's responsibility to contact this hospital to obtain all SAE relevant information and documentation.

SAEs still ongoing at EOS must be followed up for 30 days after Valchlor discontinuation or until resolution or stabilization, or until the event outcome is provided, e.g., fatal outcome.

# 7.3 Reporting of pregnancy

Any pregnancy occurring during the administration of Valchlor, including the 30 days following product discontinuation, must be reported within 24 hours or 1 working day of the investigator's knowledge of the event.

Pregnancies must be reported by the investigator on the Actelion Pregnancy Form, which is faxed or forwarded via the above-mentioned Actelion US Drug Safety email addresses within 24 hours of the investigator's knowledge of the event.

Any pregnancy diagnosed in the female partner of a male subject during treatment with Valchlor must be reported to Actelion US Drug Safety within 24 hours of the investigator's knowledge of the event.

Epidemiology and Observational Studies AC-079A501 Version 3


# 7.3.1 Follow-up of pregnancy

If subsequent follow-up information is required, Actelion US Drug Safety will send a DCF directly to the investigator.

Any pregnancy must be followed to its conclusion and its outcome must be reported to Actelion US Drug Safety directly.

# 7.4 Reconciliation

Actelion Operations (Clinical Study Leader) will keep a tracking log of all SAEs sent to Actelion US Drug Safety and the corresponding Actelion acknowledgement of receipt with Actelion MCN, so that reconciliation can be performed either periodically and/or at the end of the non-interventional study.

# 8 PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS

The Scientific Committee, in collaboration with Actelion, will publish data from this study at conferences and in journals when the sample size for analyses is sufficient.

# 9 DATA OWNERSHIP

Actelion Pharmaceuticals US, Inc. owns the data.

# 10 STUDY COMMITTEE(S)

An independent Scientific Committee of 4–6 key opinion leaders in the field of MF-CTCL has been appointed and their responsibilities will provide scientific input on the MF-CTCL Study protocol and review of study data.


### 11 REFERENCES


- [Agar 2010] Agar NS, Wedgeworth E, Crichton S, et al. Survival outcomes and prognostic factors in mycosis fungoides/Sezary syndrome: validation of the revised International Society for Cutaneous Lymphomas/European Organisation for Research and Treatment of Cancer staging proposal. J Clin Oncol. 2010;28(31):4730–39.
- [Chren 1996] Chren MM, Lasek RJ, Quinn LM, Mostow EN, Zyzanski SJ. Skindex, a quality-of-life measure for patients with skin disease: reliability, validity and responsiveness. J Invest Dermatol. 1996 Nov;107(5):707-13.
- [Chren 1997a] Chren MM, Lasek RJ, Quinn LM, Covinsky KE. Convergent and discriminant validity of a generic and a disease-specific instrument to measure quality of life in patients with skin disease. J Invest Dermatol. 1997;108(1):103–07.
- [Chren 1997b] Chren MM, Lasek RJ, Flock SA, Zyzanski SJ. Improved discriminative and evaluative capability of a refined version of skindex, a quality-of-life instrument for patients with skin diseases. Arch Dermatol. 1997;133:1433,1440.
- [Chren 2001] Chren MM, Lasek RJ, Sahay AP, Sands LP. Measurement of properties of skindex-16, a brief quality-of-life measure for patients with skin diseases. J Cutan Med Surg. 2001 Mar-Apr;5(2):105-10. Epub 2001 Mar 21.
- [Criscione 2007] Criscione VD, Weinstock MA. Incidence of cutaneous T-cell lymphoma in the United States, 1973–2002. Arch Dermatol. 2007;143(7):854–859.
- [Imam 2013] Imam MH, Shenoy PJ, Flowers CR, Phillips A, Lechowicz MJ. Incidence and survival patterns of cutaneous T-cell lymphomas in the United States. Leuk Lymphoma. 2013;54(4):752–9.
- [Kim 2003a] Kim YH, Liu HL, Mraz-Gernhard S, Varghese A, Hoppe RT. Long-term outcome of 525 patients with mycosis fungoides and Sezary syndrome: clinical prognostic factors and risk for disease progression. Arch Dermatol. Jul 2003;139(7):857–66.
- [Kim 2003b] Kim YH, Martinez G, Varghese A, Hoppe RT. Topical nitrogen mustard in the management of mycosis fungoides: update of the Stanford experience. Arch Dermatol. 2003;139(2):165–73.
- [Kim 2014] Kim EE, Duvic M, Guitart J, Lessin S. Efficacy and safety of mechlorethamine (MCH) 0.04% gel in mycosis fungoides (MF) after treatment with topical MCH 0.02%. Presented at the American Society of Clinical Oncology (ASCO) 50<sup>th</sup> Annual Meeting. Chicago, IL. May 30–Jun 3 2014. Poster #9093. http://meetinglibrary.asco.org.


IF-CTCL Doc No D-16.626


- [Korgavkar 2013] Korgavkar K, Xiong M, Weinstock M. Changing incidence trends of cutaneous T-cell lymphoma. JAMA Dermatol. 2013;149(11):1295–1299.
- [Lessin 2013] Lessin SR, Duvic M, Guitart J, et al. Topical chemotherapy in cutaneous T-cell lymphoma: positive results of a randomized, controlled, multicenter trial testing the efficacy and safety of a novel mechlorethamine, 0.02%, gel in mycosis fungoides. JAMA Dermatol. 2013;149(1):25–32.
- [Leukemia & Lymphoma Society 2011] Leukemia & Lymphoma Society [Internet] Cutaneous T-Cell Lymphoma Facts 2011 [accessed 22 October 2014]. Available from:
  - http://www.lls.org/#/resourcecenter/freeeducationmaterials/lymphoma/cutaneoustcell.
- [Lymphoma.org 2011] Lymphoma Research Foundation. [Internet] Cutaneous T-cell lymphoma: Types of Cutaneous T-Cell Lymphoma [accessed 22 October 2014]. Available from: http://www.lymphoma.org/site/pp.asp?c=bkLTKaOQLmK8E&b=6300151.
- [NCCN 2014] National Comprehensive Cancer Network Clinical Practice Guidelines in Oncology: Non-Hodgkin's Lymphomas. Version 4 .2014 [accessed on 22 August 2014]. Available from: http://www.nccn.org/professionals/physician\_gls/pdf/nhl.pdf.
- [PatientsLikeMe 2016] Creation of the Cutaneous T-cell Lymphoma-Quality of Life (CTCL-QoL) measure. Actelion Pharmaceuticals Ltd. Final Report. 31 May 2016.
- [Ramsay 1995] Ramsay DL, Meller JA, Zackheim HS. Topical treatment of early cutaneous T-cell lymphoma. Hematol Oncol Clin North Am. 1995;9(5):1031–56.
- [Reich 2012] Reich A, Heisig M, Phan NQ, et al. Visual analogue scale: evaluation of the instrument for the assessment of pruritus. Acta Derm Venereol. 2012;92(5): 497–501.
- [Scarisbrick 2014] Scarisbrick JJ, Kim YH, Whittaker SJ, et al. Prognostic Factors, Prognostic Indices and Staging in Mycosis Fungoides and Sezary Syndrome: Where are we now? Br J Dermatol 2014 Jun;170(6):1226–36.


Doc No D-16.626


# Appendix A Skindex-29 Questionnaire

Skindex29 ©MMChren,1996

These questions concern your feelings over the past 4 weeks about **the skin condition that has bothered you the most**. Check the answer that comes closest to the way you have been feeling.

| HOW OFTEN DURING THE PAST FOUR WEEKS DO THESE STATEMENTS DESCRIBE YOU? | NEVER | RARELY | SOMETIMES | OFTEN | ALL THE |
|---|---|---|---|---|---|
| 1. My skin hurts | | □₂ | □₃ | □₄ | □₅ |
| 2. My skin condition affects how well I sleep | | | □₃ | □₄ | □₅ |
| 3. I worry that my skin condition may be serious | | | □₃ | □₄ | □₅ |
| 4. My skin condition makes it hard to work or do hobbies | | | □₃ | □₄ | □₅ |
| 5. My skin condition affects my social life | | | □₃ | □₄ | □₅ |
| 6. My skin condition makes me feel depressed | | | □₃ | □₄ | □5 |
| 7. My skin condition burns or stings | | | □₃ | □₄ | □₅ |
| 8. I tend to stay at home because of my skin condition | | | □₃ | □₄ | □₅ |
| 9. I worry about getting scars from my skin condition | | | □₃ | □₄ | □₅ |
| 10. My skin itches | | | □₃ | □₄ | □₅ |
| 11. My skin condition affects how close I can be with those I love . | | | □₃ | □₄ | □5 |
| 12. I am ashamed of my skin condition | | | □₃ | □₄ | □₅ |
| 13. I worry that my skin condition may get worse | | | □₃ | □4 | □₅ |
| 14. I tend to do things by myself because of my skin condition . | | | □₃ | □₄ | □₅ |
| 15. I am angry about my skin condition | | | □₃ | □₄ | □₅ |
| 16. Water bothers my skin condition (bathing, washing hands) . | | | □₃ | □₄ | □₅ |
| 17. My skin condition makes showing affection difficult | | | □₃ | □₄ | □5 |
| 18. I worry about side-effects from skin medications / treatments . | | | □₃ | □₄ | □₅ |
| 19. My skin is irritated | | | □₃ | □₄ | □₅ |
| 20. My skin condition affects my interactions with others | | □₂ | □₃ | □₄ | □5 |

Please turn to next page

Skindex29 – United States/English – Original version 8kindex29\_AU2.0\_eng-U8orl.doc


Skindex29 ©MMChren,1996


These questions concern your feelings over the past 4 week about **the skin condition that has bothered you the most**. Check the answer that comes closest to the way you have been feeling.

| HOW OFTEN DURINGTHE PAST 4 WEEK<br>DO THESE STATEMENTS DESCRIBE YOU? | | RARELY | SOMETIMES | OFTEN | ALL THE<br>TIME |
|---|---|---|---|---|---|
| 21. I am embarrassed by my skin condition | <b>□</b> ₁ | □₂ | □₃ | □₄ | □₅ |
| 22. My skin condition is a problem for the people I love | | | □₃ | □₄ | □₅ |
| 23. I am frustrated by my skin condition | | | □₃ | □₄ | □₅ |
| 24. My skin is sensitive | | | □₃ | □₄ | □₅ |
| 25. My skin condition affects my desire to be with people | | | □₃ | □₄ | □₅ |
| 26. I am humiliated by my skin condition | | | □₃ | □₄ | □₅ |
| 27. My skin condition bleeds | | | □₃ | □₄ | □₅ |
| 28. I am annoyed by my skin condition | | | □₃ | □₄ | □₅ |
| 29. My skin condition interferes with my sex life | | | □₃ | □₄ | □₅ |
| 30 My skin condition makes me tired | | | □₃ | □₄ | <b>□</b> ₅ |

# AC-079A501 Version 3


#### **Skindex-29 Scoring algorithm** Appendix B



Scaling and Scoring Version 2.0: February 2012


# **Domains and Clusters**

### Skindex-29:

| Domains | Number of<br>Items | Cluster of<br>Items | Item<br>reversion | Direction of Domains |
|---|---|---|---|---|
| Emotions | 10 | 3; 6; 9; 12;<br>13; 15; 21;<br>23; 26; 28 | | |
| Symptoms | 7 | 1; 7; 10; 16;<br>19; 24; 27 | No | Higher score = higher impact of skin disease |
| Functioning | 12 | 2; 4; 5; 8; 11;<br>14; 17; 20;<br>22; 25; 29; 30 | | |

# **Scoring of Domains**

# Skindex-29:

| Item scaling | 5-point Likert-type scale |
|---|---|
| Weighting of items | No |
| Range of scores | From 0 (no effect) to 100 (effect experienced all the time) |
| Scoring Procedure | All responses are transformed to a linear scale of 100. Transformed item scores: never = 0 rarely = 25 sometimes = 50 often = 75 all the time = 100 Scale scores: A scale score is the mean of a patient's responses to the items in a given scale. Note: Item 18 is a single item, not included in scoring. |

| Interpretation and<br>Analysis of missing<br>data | <ul> <li>If responses to more than 25% of items are missing overall, the questionnaire is eliminated.</li> <li>If any scale has more than 25% of the responses missing, the scale is missing.</li> <li>Scale scores are the average of non-missing items in a given scale.</li> </ul> |
|---|---|
| Interpretation of multiple answers for one item | An item with multiple answers is considered missing. |

Copyright © 2012 Mapi Research Trust-All rights reserved

Doc No D-16.626

AC-079A501 Version 3


# Appendix C Visual Analog Scale for pruritus




IF-CTCL Doc No D-16.626


# Appendix D Mycosis fungoides/Sézary syndrome-type cutaneous T-cell lymphoma

# The CTCL-QoL Final Version

Please complete these items regarding your experiences over the past 4 weeks.

| In the past 4 weel | īs | | | |
|---|---|---|---|---|
| Q1how much did | you worry that your my | cosis fungoides or Séza | ry syndrome may g | et worse? |
| 1 | 2 | 3 | 4 | 5 |
| Not at all | A little bit | Somewhat | Quite a bit | Very much |
| Q2how often did | you feel hopeless becau | se of having mycosis fu | ngoides or Sézary s | yndrome? |
| 1 | 2 | 3 | 4 | 5 |
| Never | Rarely | Sometimes | Often | Always |
| Q3how frustrates | l were you by the unpre | dictability of mycosis fu | ngoides or Sézary s | yndrome? |
| l I | 2 | 3 | 4 | 5 |
| Not at all | A little bit | Somewhat | Quite a bit | Very much |
| Q4how often did y | ou feel depressed or sad | l because of mycosis fur | rgoides or Sézary sy | ndrome? |
| 1 | 2 | 3 | 4 | 5 |
| Never | Rarely | Sometimes | Often | Always |
| 05how confident | lid yo u feel about mana | ging vour mycosis fung | oides or Sézarv syn | |
| 1 | 2 | 3 | 4 | 5 |
| Absolutely confiden | t Very confident | Moderately 1 | Mildly confident | Not at all |
| Troscialci, comina | t very community | confident | andly confident | confident |
| O6 how severe we | re your mycosis fungoi | | читане? | |
| 1 | 7 | 3 4 | 5 | Does not apply (I |
| Not at all Al | ittle severe Somew | hat severe Severe | Very severe | don't have |
| Tional and Tra | ittle severe bomew. | man severe bevere | very severe | symptoms right |
| | | | | now) |
| O7 how hardows | ome was your mycosis f | ungoides or Cézani mud | vom a traa tmant? | |
| 1 | nie nes your mycosis ji | A STANSON OF THE PARTY SPILLS | 5 | Does not apply (I |
| Not at all | A little Some | 1 | - | |
| | | | Very | don't have |
| | rdensome burden | | Very<br>Burdensome | symptoms right |
| burdensome bu | rdensome burden | some | Burdensome | symptoms right<br>now) |
| Durdensome bu Q8how much did | irdensome burden<br>lyour mycosis fungoide | some<br>s <i>or Sézary syndrome lin</i> | Burdensome<br>nityour daily activ | symptoms right<br>now) |
| Durdensome bu Q8how much did | rdensome burden | some<br>s <i>or Sézary syndrome lin</i> | Burdensome<br>nityour daily activ | symptoms right<br>now) |
| Q8how much did<br>and outside of the h | rdensome burden<br>Lyour mycosis fungoide<br>ouse, self-care such as c<br>2 | some<br>g <i>or Sézary syndrome lin</i><br>cooking, cleaning, gettin<br>3 | Burdensome<br>nit your daily activing dressed, etc.)?<br>4 | symptoms right<br>now)<br>ties (work inside |
| Q8how much did<br>and outside of the h<br>l<br>Not at all | rdensome burden<br>Lyour mycosis fungoide<br>ouse, self-care such as c<br>2<br>A little bit | some<br>g <i>or Sézary syndrome lin<br/>cooking, cleaning, gettin</i><br>3<br>Somewhat | Burdensome nityour daily activity ag dressed, etc.)? 4 Quite a bit | symptoms right now) thes (work inside 5 Very much |
| Q8how much did<br>and outside of the h<br>l<br>Not at all<br>Q9how often did | lyour mycosis fungoide<br>ouse, self-care such as c<br>2<br>A little bit<br>mycosis fungoides or Se | some<br>g <i>or Sézary syndrome lin<br/>cooking, cleaning, gettin</i><br>3<br>Somewhat | Burdensome nityour daily activity ag dressed, etc.)? 4 Quite a bit | symptoms right now) thes (work inside 5 Very much |
| Q8how much did<br>and outside of the h<br>l<br>Not at all<br>Q9how often did | rdensome burden<br>Lyour mycosis fungoide<br>ouse, self-care such as c<br>2<br>A little bit | some<br>g <i>or Sézary syndrome lin<br/>cooking, cleaning, gettin</i><br>3<br>Somewhat | Burdensome nityour daily activity ag dressed, etc.)? 4 Quite a bit | symptoms right now) thes (work inside 5 Very much |
| Q8how much did and outside of the h Not at all Q9how often did you too tired to work | lyour mycosis fungoide<br>ouse, self-care such as c<br>2<br>A little bit<br>mycosis fungoides or Se | some sor Sézary syndrome lin cooking, cleaning, gettin 3 Somewhat ézary syndrome (the con | Burdensome nit your daily activity ng dressed, etc.)? 4 Quite a bit ndition or associated | symptoms right now) thes (work inside 5 Very much |
| Q8how much did<br>and outside of the h<br>l<br>Not at all<br>Q9how often did | lyour mycosis fungoide<br>ouse, self-care such as c<br>2<br>A little bit<br>mycosis fungoides or Se | some<br>g <i>or Sézary syndrome lin<br/>cooking, cleaning, gettin</i><br>3<br>Somewhat | Burdensome nityour daily activity ag dressed, etc.)? 4 Quite a bit | symptoms right now) thes (work inside 5 Very much |
| Q8how much did and outside of the h l Not at all Q9how often did you too tired to work l Never | lyour mycosis fungoide<br>ouse, self-care such as c<br>2<br>A little bit<br>mycosis fungoides or Se<br>k or do daily activities? | some or Sézary syndrome lin cooking, cleaning, gettin 3 Somewhat ézary syndrome (the con 3 Sometimes | Burdensome nityour daily activity ng dressed, etc.)? 4 Quite a bit udition or associated 4 Often | symptoms right now) ties (work inside 5 Very much d treatment) leave 5 Always |
| Q8how much did and outside of the h l Not at all Q9how often did you too tired to work l Never | lyour mycosis fungoides ouse, self-care such as c 2 A little bit mycosis fungoides or Se k or do daily activities? 2 Rarely d mycosis fungoides or | some or Sézary syndrome lin cooking, cleaning, gettin 3 Somewhat ézary syndrome (the con 3 Sometimes | Burdensome nityour daily activity ng dressed, etc.)? 4 Quite a bit udition or associated 4 Often | symptoms right now) ties (work inside 5 Very much d treatment) leave 5 Always |
| Q8how much did and outside of the h l Not at all Q9how often did you too tired to work l Never Q10how much did | lyour mycosis fungoides ouse, self-care such as c 2 A little bit mycosis fungoides or Se k or do daily activities? 2 Rarely d mycosis fungoides or | some or Sézary syndrome lin cooking, cleaning, gettin 3 Somewhat ézary syndrome (the con 3 Sometimes | Burdensome nityour daily activity ng dressed, etc.)? 4 Quite a bit udition or associated 4 Often | symptoms right now) ties (work inside 5 Very much d treatment) leave 5 Always |
| Q8how much did and outside of the h 1 Not at all Q9how often did you too tired to work 1 Never Q10how much did others close to you? | lyour mycosis fungoides ouse, self-care such as o 2 A little bit mycosis fungoides or Se k or do daily activities? 2 Rarely d mycosis fungoides or | some g or Sézary syndrome lir cooking, cleaning, gettin 3 Somewhat ézary syndrome (the con 3 Sometimes Sézary syndrome negati | Burdensome nityour daily activity of dressed, etc.)? 4 Quite a bit idition or associated 4 Often ively affect your reli | symptoms right now) thes (work inside 5 Very much directment) leave 5 Always ationships with |
| Durdensome bu Q8how much did and outside of the hi Not at all Q9how often did you too tired to work Never Q10how much di others close to you? Not at all | lyour mycosis fungoides ouse, self-care such as o 2 A little bit mycosis fungoides or Se k or do daily activities? 2 Rarely d mycosis fungoides or 2 A little bit | some sor Sézary syndrome lin cooking, cleaning, gettin 3 Somewhat ézary syndrome (the con 3 Sometimes Sézary syndrome negati | Burdensome nityour daily activity dressed, etc.)? 4 Quite a bit udition or associated 4 Often wely affect your rel 4 Quite a bit | symptoms right now) ities (work inside 5 Very much direatment) leave 5 Always ationships with 5 Very much |
| Durdensome bu Q8how much did and outside of the hi Not at all Q9how often did you too tired to work I Never Q10how much di others close to you? I Not at all Q11how often did | lyour mycosis fungoides ouse, self-care such as o 2 A little bit mycosis fungoides or Se k or do daily activities? 2 Rarely d mycosis fungoides or 2 A little bit dyou feel that others do | some sor Sézary syndrome lin cooking, cleaning, gettin 3 Somewhat ézary syndrome (the con 3 Sometimes Sézary syndrome negati | Burdensome nityour daily activity dressed, etc.)? 4 Quite a bit udition or associated 4 Often wely affect your rel 4 Quite a bit | symptoms right now) ities (work inside 5 Very much direatment) leave 5 Always ationships with 5 Very much |
| Durdensome bu Q8how much did and outside of the hi Not at all Q9how often did you too tired to work Never Q10how much di others close to you? Not at all | lyour mycosis fungoides ouse, self-care such as o 2 A little bit mycosis fungoides or Se k or do daily activities? 2 Rarely d mycosis fungoides or 2 A little bit dyou feel that others do | some sor Sézary syndrome lin cooking, cleaning, gettin 3 Somewhat ézary syndrome (the con 3 Sometimes Sézary syndrome negati | Burdensome nityour daily activity dressed, etc.)? 4 Quite a bit udition or associated 4 Often wely affect your rel 4 Quite a bit | symptoms right now) ities (work inside 5 Very much direatment) leave 5 Always ationships with 5 Very much |
| Durdensome bu Q8how much did and outside of the hi Not at all Q9how often did you too tired to work I Never Q10how much di others close to you? I Not at all Q11how often dif fungoides or Sézary | lyour mycosis fungoides ouse, self-care such as o 2 A little bit mycosis fungoides or Se k or do daily activities? 2 Rarely id mycosis fungoides or 4 A little bit dyou feel that others do syndrome? 2 | some sor Sézary syndrome lin cooking, cleaning, gettin 3 Somewhat izary syndrome (the con 3 Sometimes Sézary syndrome negati 3 Somewhat not understand what ye | Burdensome nityour daily activity of daily of da | symptoms right now) ties (work inside 5 Very much direatment) leave 5 Always ationships with 5 Very much gh with mycosis |
| burdensome bu Q8how much did and outside of the hi Not at all Q9how often did you too tired to work 1 Never Q10how much did others close to you? 1 Not at all Q11how often did fungoides or Sécary 1 Never | lyour mycosis fungoides ouse, self-care such as o A little bit mycosis fungoides or Se k or do daily activities? 2 Rarely d mycosis fungoides or 2 A little bit dyou feel that others do syndrome? 2 Rarely | some sor Sézary syndrome lin cooking, cleaning, gettin 3 Somewhat zary syndrome (the con 3 Sometimes Sézary syndrome negati 3 Somewhat not understand what you | Burdensome nityour daily activity dressed, etc.)? 4 Quite a bit dition or associated 4 Often wely affect your rel 4 Quite a bit ou are going throug 4 Often | symptoms right now) ties (work inside 5 Very much direatment) leave 5 Always ationships with 5 Very much the with mycosis Always |
| Durdensome bu Q8how much dia and outside of the hi Not at all Q9how often did you too tired to work I Never Q10how much di others close to you? I Not at all Q11how often di fungoides or Sézary I Never Q12 to what exter | lyour mycosis fungoides ouse, self-care such as o 2 A little bit mycosis fungoides or Se k or do daily accivities? 2 Rarely id mycosis fungoides or 2 A little bit dyou feel that others do syndrome? 2 Rarely ut did mycosis fungoides | some sor Sézary syndrome lin cooking, cleaning, gettin 3 Somewhat zary syndrome (the con 3 Sometimes Sézary syndrome negati 3 Somewhat not understand what you 3 Sometimes cor Sézary syndrome me | Burdensome nityour daily activity dressed, etc.)? 4 Quite a bit dition or associated 4 Often wely affect your rel 4 Quite a bit ou are going throug 4 Often | symptoms right now) ties (work inside 5 Very much direatment) leave 5 Always ationships with 5 Very much the with mycosis Always |
| Durdensome bu Q8how much dia and outside of the hi Not at all Q9how often did you too tired to work I Never Q10how much di others close to you? I Not at all Q11how often di fungoides or Sézary I Never Q12 to what exter | lyour mycosis fungoides ouse, self-care such as o A little bit mycosis fungoides or Se k or do daily activities? 2 Rarely d mycosis fungoides or 2 A little bit dyou feel that others do syndrome? 2 Rarely | some sor Sézary syndrome lin cooking, cleaning, gettin 3 Somewhat zary syndrome (the con 3 Sometimes Sézary syndrome negati 3 Somewhat not understand what you 3 Sometimes cor Sézary syndrome me | Burdensome nityour daily activity dressed, etc.)? 4 Quite a bit dition or associated 4 Often wely affect your rel 4 Quite a bit ou are going throug 4 Often | symptoms right now) ties (work inside 5 Very much direatment) leave 5 Always ationships with 5 Very much the with mycosis Always |
| Durdensome bu Q8how much dia and outside of the hi Not at all Q9how often did you too tired to work I Never Q10how much di others close to you? I Not at all Q11how often di fungoides or Sézary I Never Q12 to what exter | lyour mycosis fungoides ouse, self-care such as o 2 A little bit mycosis fungoides or Se k or do daily accivities? 2 Rarely id mycosis fungoides or 2 A little bit dyou feel that others do syndrome? 2 Rarely ut did mycosis fungoides | some sor Sézary syndrome lin cooking, cleaning, gettin 3 Somewhat zary syndrome (the con 3 Sometimes Sézary syndrome negati 3 Somewhat not understand what you 3 Sometimes cor Sézary syndrome me | Burdensome nityour daily activity dressed, etc.)? 4 Quite a bit dition or associated 4 Often wely affect your rel 4 Quite a bit ou are going throug 4 Often | symptoms right now) ties (work inside 5 Very much direatment) leave 5 Always ationships with 5 Very much the with mycosis Always |


# Appendix E Mycosis fungoides/Sézary syndrome-type cutaneous T-cell lymphoma (CTCL QOL Scoring)

Scoring the CTCL-QoL

A total raw CTCL-QoL score is calculated by adding up the patient's total score from the 12 CTCL-QoL items. The Raw to Scaled Score Conversion Table provides scaled scores (M = 100, SD = 15) that correspond to the CTCL-QoL total score. Although total raw scores of 10 or 11 are possible due to two items with the response choice "Does not apply (I don't have symptoms right now)", these scores should not be interpreted differently from a score of 12. For scoring purposes, "Does not apply (I don't have symptoms right now)" is scored as a 0. Further, in order to score the CTCL-QoL, each of the 12 items must be completed.

Raw to Scaled Score Conversion Table

| and the contract of the contract | Raw CTCL-QoL | | |
|---|---|---|---|
| Raw CTCL-QoL Score | Scaled Score | Score, Continued | Scaled Score |
| 12 or below | 62 | 37 | 113 |
| 13 | 74 | 38 | 114 |
| 14 | 80 | 39 | 115 |
| 15 | 84 | 40 | 116 |
| 16 | 87 | 41 | 117 |
| 17 | 89 | 42 | 118 |
| 18 | 91 | 43 | 119 |
| 19 | 93 | 44 | 120 |
| 20 | 94 | 45 | 121 |
| 21 | 96 | 46 | 123 |
| 22 | 97 | 47 | 124 |
| 23 | 98 | 48 | 125 |
| 24 | 100 | 49 | 126 |
| 25 | 101 | 50 | 128 |
| 26 | 102 | 51 | 129 |
| 27 | 103 | 52 | 131 |
| 28 | 104 | 53 | 133 |
| 29 | 105 | 54 | 135 |
| 30 | 106 | 55 | 137 |
| 31 | 107 | 56 | 139 |
| 32 | 108 | 57 | 143 |
| 33 | 109 | 58 | 147 |
| 34 | 110 | 59 to 60 | 154 |
| 35 | 111 | | |
| 36 | 112 | | |

<sup>&</sup>lt;sup>1</sup> Scaled scores were standardized on the current sample to have a mean of 100 and a standard deviation of 15

<sup>&</sup>lt;sup>2</sup> While it is possible to obtain a raw score of 10 or 11 due to endorsing "Does not apply (I don't have symptoms right now)" to CTCL-QoL items, these scores should be viewed as equivalent to a 12.